CLINICAL TRIAL: NCT04048525
Title: Cytokine Removal With CVVHD Using a Membrane With Adsorption Capacity: A Pilot Randomized Trial
Brief Title: Cytokine Removal With CVVHD Compared to CVVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, JOSE LUIS PEREZ FERNANDEZ, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CYTOHUB
Record Dates: First submitted 2019-02-13; First posted 2019-08-07 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2019-08

CONDITIONS: Cytokine Release Syndrome; Sepsis; AKI
Keywords: CRRT; CVVHD; CVVH
MeSH Terms: conditions — Cytokine Release Syndrome; Sepsis | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVVHD with ST150 (Experimental): Patients with sepsis whom present AKI meeting CRRT initiation criteria will be started on CVVHD with PrismafleX eXeed™ II (Hospal) using an ST150SET copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface. Anticoagulation of the ST150 set with unfractioned heparin will only be initiated if there´s no clinical contraindication. ST150 set will be changed when clotted and every 24 hours during the first 72 hours of CVVHD. No citrate anticoagulation will be used.
  Interventions: Procedure: CVVHD
- CVVH with ST150 (Active Comparator): Patients with sepsis whom present AKI meeting CRRT initiation criteria will be started on CVVH with PrismafleX eXeed™ II (Hospal) using an ST150SET copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface. Anticoagulation of the ST150 set with unfractioned heparin will only be initiated if there´s no clinical contraindication. ST150 set will be changed when clotted and every 24 hours during the first 72 hours of CVVH. No citrate anticoagulation will be used.
  Interventions: Procedure: CVVH

INTERVENTIONS:
Procedure: CVVHD — CVVHD will be used during 72 hours with a prescribed dose of 30 ml/Kg/h Prismasol® 4 as dialysate fluid. Blood flow of 200-250 ml/min, to achieve 12 - 15 L/h will be prescribed. Isovolemic CRRT will be encouraged during this 72 hours if volume overload status is not present. After 72 hours, CVVHD will be continued and dialysate dose (ml/kg/h) will be adjusted to achieve creatinine levels between 80-120 umol/L until patient recovers urine output and / or tolerates intermittent hemodialysis.
  Other Names: Continuous venovenous hemodialysis
  Arms: CVVHD with ST150
Procedure: CVVH — CVVH will be used during 72 hours with a prescribed dose of 30 ml/Kg/h Prismasol® 4 as reposition fluid. Blood flow of 200-250 ml/min, to achieve 12 - 15 L/h will be prescribed adjusting the adequate percentage of prefilter infusion to maintain a theoretical filtration fraction between 18-22%. Isovolemic CRRT will be encouraged if volume overload status is not present. After 72 hours, CVVH will be continued and filtration dose (ml/kg/h) will be adjusted to achieve creatinine levels between 80-120 umol/L until patient recovers urine output and / or tolerates intermittent hemodialysis.
  Other Names: Continuous venovenous haemofiltration
  Arms: CVVH with ST150

SUMMARY:
Septic patients with acute kidney injury (SA-AKI) requiring continuous renal replacement therapies (CRRT) present high mortality due to systemic inflammatory response, cytokine liberation, and finally multiorgan dysfunction. Cytokine plasmatic elimination with continuous venovenous hemofiltration (CVVH) presents a high resource cost both technical and human. The study primary end-point is to demonstrate a similar cytokine removal of continuous venovenous hemodialysis (CVVHD) respect to CVVH, both modalities employing the same adsorption capacity membrane. As secondary end-points investigators will try to demonstrate technical superiority of CVVHD respect to CVVH. In order to achieve these objectives investigators have designed a proof of concept exploratory trial that will include those participants whom present SA-AKI meeting CRRT initiation criteria. During the first 72 hours investigators will measure plasmatic elimination capacity of main cytokines, and other clinical and prognostic relevant molecules. Investigators wil measure mean filter life during all CRRT with special attention to the first 72 hours. Investigators will also measure hemodynamic, respiratory, and metabolic parameters. Finally, investigators will analyze 90 days survival. Demonstration of a similar immunomodulating capacity and a minor complication rate with its consequent lower cost, should settle the based evidence principles that recommend the use of CVVHD associated to an adsorption capacity membrane in patients with SA-AKI whom need CRRT.

DETAILED DESCRIPTION:
Investigators will warrant a correct protocol application. Study data will be reviewed by an external monitoring committee from the clinical assay research central unit (UCICEC - IDIBELL). Monitors will contrast registered data from the collection data form (CDF) with data from patient´s medical record. All patient´s medical records will be indefinitely saved in electronical format to be reviewed if necessary. Participants who meet inclusion criteria will be randomized for one of both arms with aleatory assignation using a randomisation sequential (RndSeq) program for Statistical Package for the Social Sciences (SPSS). Investigators will report adverse events (in less than 24 hours if severe) to the sponsor center to be properly evaluated. If the severe adverse event (SAE) is finally evaluated by the study board as related to the intervention arm, urgent notification to health authorities must proceed and study should be interrupted until further decision. Data registry has been created to include all variables with written individual data collection forms (DCF). Data will be bedside registered by the investigators but final software database registration will be done by the statistics outside investigator who has no contact with the participant situation. Cytokines levels will be introduced in DCF when measured (every six months). Statistical analysis will be done by the statistics investigator who wont have any role in patient´s selection, randomization, or follow up. SPSS v. 18.0 for statistical analysis will be used. Variable distribution will be studied and logarithmic transformation will be used on those variables that don't present normal distribution, presumably cytokine levels. Univariate analysis comparing clinical, demographic, biochemical, metabolic, hemodynamic and respiratory baseline variables between both arms (CVVHD and CVVH), will be done with two-tailed t test for continuous variables and chi-square test for categorical variables. Variables determined several times (T0, T24, T48, T72) will be analysed using a one-way repeated measures ANOVA test in order to demonstrate differences between both arms. Multivariate analysis will be completed to control those clinically relevant confounding variables as well as to discover baseline differences. According to hypothesis and to the dependent variable on study, investigators will use a survival analysis (to study mortality) with a cox regression model, or a hierarchic multiple linear regression model when the dependent variable is continuous. Arm intervention (CVVHD, CVVH) will be considered as the main independent variable adding other control independent variables. As the study is measuring cytokine levels in five different moments (T0, T24, T48, T72), in order to maximize statistical power and reduce control variables number, the area under the curve (AUC) we´ll be determined for every cytokine during the first 72 hours. Due to this statistical maneuver, investigators will obtain a continuous variable that represents each cytokine level during the biochemical study period (72 hours). To evaluate if the arm intervention improvement in terms of efficacy and safety could be related to cytokine levels during the first 72 hours, a mediation complementary analysis will be done considering cytokine (represented by AUC) as a mediator between the independent variable (intervention arm) and the evaluated effect.

ELIGIBILITY:
Inclusion Criteria:

* Less than 72 hours from ICU admission to inclusion
* Clinical diagnosis of Severe Sepsis or Septic shock (SCCM definitions)
* Correct therapeutic initial management of septic process (SSC guidelines)
* Clinical diagnosis of Acute Kidney Injury (ADQI definitions)
* Acute Kidney Injury meeting CRRT initiation criteria (ADQI guidelines)
* Written informed consent from patient or legal surrogates

Exclusion Criteria:

* End Stage Renal Disease(ESRD)
* Received previous CRRT or hemodialysis in the last three months
* Inclusion in other ongoing study
* Coexisting illness with a high probability of death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Cytokine specific removal (0-72h) | 72 hours
  Cytokine concentration changes between baseline and 72 hours for each cytokine: interleukin-1β (IL-1β), tumor necrosis factor α (TNF-α), interleukin 6 (IL-6), interleukin-4 (IL-4), and interleukin-10 (IL-10) levels will be determined in plasma. Changes will be expressed in percentages respect to baseline concentrations for each cytokine. Determinations should only be done when ST150 set has been working for at least 6 continuous hours. This means that determinations can be advanced or delayed +/- 4 hours to scheduled time (for example 68 - 76 hours for T72).

SECONDARY OUTCOMES:
Cardiovascular SOFA score variations. | 72 hours
  Cardiovascular SOFA score will be registered every 24 hours (0-4) and variation from baseline to 72 hours will be evaluated calculating the Delta cardiovascular SOFA score from baseline to 72 h (SUM of the 4 daily SOFA scores).
Respiratory SOFA score variations. | 72 hours
  Respiratory SOFA score (0-4) will be registered every 24 hours and variation from baseline to 72 hours will be evaluated calculating the Delta respiratory SOFA score from baseline to 72 h (SUM of the 4 daily SOFA scores).
Number of filters employed. | 72 hours
  Number of times set was changed during the first 72 hours on CRRT.
Rate of dialytrauma events | 72 hours
  Rate of adverse events related to CRRT known as "dialytrauma". Red blood cells transfusions related with filter clotting, thrombocytopenia (less than 100.000), hypophosphatemia (less than 0.7 mmol/L), hypokaliemia (less than 3.3 mmol/ L), and hypothermia (less than 35.5ºC rectal temperature).
Sieving coefficients for plasma solutes | 0-72 hours
  Sieving coefficients for plasma solutes (creatinine, urea, potassium, albumine, magnesium, phosphate, and others) will be determined after measuring blood (pre and postfilter) and ultrafiltrate levels at 24 hours, 48 hours, and 72 hours.
  24h, 48h, and 72h determinations should only be done when ST150 set has been working for at least 6 continuous hours. This means that determinations can be advanced or delayed +/- 4 hours to scheduled time (for example 20 - 28 hours for T24).
Survival at 90 days after randomization | 90 days
  Kaplan Meyer survival analysis and cox proportional hazard ratio for death will be both done at 90 days after CRRT initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ordoñez-Llanos, PhD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No